CLINICAL TRIAL: NCT06307821
Title: Assessing the Impact of Weizmannella Coagulans BC99 on Protein Digestion and Metabolism: A Randomized, Double-Blind Controlled Trial
Brief Title: the Role of Probiotic in Protein Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024002
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Probiotic; Protein digestion
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double（Participant,Investigator）
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): 48 billion CFU/day BC99 and protein powder; Storage: sealed, protected from light, placed in a cool and dry place.
  Interventions: Dietary Supplement: Probiotic
- placebo (Placebo Comparator): Protein powder, 8 bags per day; Storage: sealed, protected from light, placed in a cool and dry place.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The intervention lasts for 12 weeks, with follow-ups conducted at weeks 0, 6, and 12 to assess participants' digestion and absorption rates of dietary protein, as well as to collect fecal samples for analysis of changes in the gut microbiota.
  Arms: Probiotics
Dietary Supplement: Placebo — The intervention lasts for 12 weeks, with follow-ups conducted at weeks 0, 6, and 12 to assess participants' digestion and absorption rates of dietary protein, as well as to collect fecal samples for analysis of changes in the gut microbiota.
  Arms: placebo

SUMMARY:
This study investigates the functional effects of probiotics on athletes by administering Weizmannella coagulans BC99 for 12 weeks. It aims to assess the probiotic's influence on skeletal muscle content, athletic performance, and protein digestion and metabolism. This is achieved by monitoring changes in digestive enzymes, amino acids, body composition, and hormone levels. The research seeks to offer a theoretical foundation for optimizing athletes' training and nutrition strategies and suggests the potential of probiotics in enhancing nutrient absorption and utilization, particularly in individuals with compromised digestive capabilities.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily, in writing, and signing the informed consent form, agreeing to participate in this study;
2. Agree to abide by the protocol and study restrictions;
3. The subject is not allergic to protein products;
4. Male or female subjects aged 18 to 35 years old (including 18 and 35 years old);
5. Male subjects should weigh no less than 50 kilograms. Female subjects must weigh no less than 45 kg. Body mass index (BMI) = weight (kg)/height (m)2, body mass index is in the range of 19.0 to 24.0 kg/m2;
6. No history of hidden risks of cardiovascular and cerebrovascular diseases, hypertension, diabetes, liver/kidney function, etc. and metabolic abnormalities.

Exclusion Criteria:

1. Patients with allergies and immune deficiency;
2. Donated blood or lost a large amount of blood (≥200 mL) within 3 months before taking the trial drug;
3. Other systemic diseases, including cardiovascular disease, lung disease, liver disease, kidney disease and other serious lesions of important organs, severe metabolic diseases (diabetes, thyroid disease), severe immune system diseases; no cardiovascular and cerebrovascular diseases, hypertension , diabetes, liver/kidney function and other hidden dangers and metabolic abnormalities.
4. Drugs that affect intestinal flora (including antibacterial drugs, microecological preparations, intestinal mucosal protective agents, Chinese patent medicines, etc.) have been used continuously for more than 1 week within 1 month before screening;
5. Subjects judged by other researchers to be unfit to participate.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Digestibility and absorption of dietary protein | 12 weeks
  After probiotic intervention, calculate the changes in subjects' digestibility and absorption rate of dietary protein based on baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Science and Technology, Luoyang, Henan, China